CLINICAL TRIAL: NCT06221241
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo and Active Drug-controlled Trial to Evaluate the Efficacy and Safety of JMKX000623 in Participants With Diabetic Peripheral Neuropathic Pain
Brief Title: Evaluate the Efficacy and Safety of JMKX000623 in Participants With Diabetic Peripheral Neuropathic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMKX0623-201
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMKX000623 (Experimental): JMKX000623 for 12 weeks
  Interventions: Drug: JMKX000623; Drug: Placebo
- Pregabalin (Active Comparator): Pregabalin for 12 weeks
  Interventions: Drug: Pregabalin; Drug: Placebo
- Placebo (Placebo Comparator): placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JMKX000623 — tablets for oral administration.
  Arms: JMKX000623
Drug: Pregabalin — capsules for oral administration.
  Arms: Pregabalin
Drug: Placebo — matched to JMKX000623 and Pregabalin

SUMMARY:
A Phase 2, Multicenter, Randomized, Double-blind, Placebo and Active Drug-controlled Trial to Evaluate the Efficacy and Safety of JMKX000623 in Participants with Diabetic Peripheral Neuropathic Pain

DETAILED DESCRIPTION:
Evaluate the Efficacy and Safety of JMKX000623 in Participants with Diabetic Peripheral Neuropathic Pain

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the procedures of this trial and provide written informed consent voluntarily;
2. Age ≥ 18 years, male or female;
3. Diagnosed with Diabetic Peripheral Neuropathic Pain for ≥ 24 weeks;
4. Visual Analog Scale (VAS) of 40-90 mm, and ADPS of 4-9;
5. HbA1c ≤ 9.0% and on a stable antidiabetic medication regimen for ≥ 4 weeks.

Exclusion Criteria:

1. With other peripheral neuropathies or painful diseases except for Diabetic Peripheral Neuropathic Pain;
2. Possibly allergic to the active ingredients or excipients of JMKX000623, pregabalin and acetaminophen, or history of ≥ 3 allergens, or with ongoing allergic conditions;
3. Received analgesic medications within 4 weeks prior to screening, or scheduled to use other analgesic medications during the trial;
4. Known treatment failure on pregabalin or gabapentin;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of the Average Daily Pain Score (ADPS) from baseline to Week 12. [ADPS is the weekly average pain score based on the 11-point numeric rating scale (NRS)] | baseline，Week 12
  Numeric Rating Scales(NRS )was a 11-point numeric rating scale ( 0[no pain] to 10 [worst possible pain]

SECONDARY OUTCOMES:
Change of the Average Daily Pain Score (ADPS) from baseline to Week 5. [ADPS is the weekly average pain score based on the 11-point numeric rating scale (NRS)] | baseline，Week 5
  Numeric Rating Scales(NRS )was a 11-point numeric rating scale ( 0[no pain] to 10 [worst possible pain]
Adverse Events | baseline，Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No